CLINICAL TRIAL: NCT00292188
Title: A 9 Week, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Study Of Pregabalin (BID) In Subject With Posttraumatic Peripheral Neuropathic Pain
Brief Title: P4 (Pregabalin for Peripheral Posttraumatic Pain)
Acronym: P4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081064
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Results first posted 2009-10-05 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2011-04

CONDITIONS: Neuralgia
Keywords: Phase 4, post-traumatic neuropathic pain, neuropathic pain, Nep, post surgical pain, nerve injury, phantom limb pain, international
MeSH Terms: conditions — Neuralgia; Pain, Postoperative; Phantom Limb | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin — pregabalin
  Arms: Active
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of pregabalin compared to placebo in the treatment of posttraumatic peripheral neuropathic pain

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Posttraumatic Peripheral Neuropathic Pain (NeP) syndrome, including post-surgical NeP, NeP due to peripheral nerve injury, and phantom limb pain, confirmed by a qualified pain specialist and persisting for a minimum of 3 months following the traumatic event

Exclusion Criteria:

* Subjects whose posttraumatic neuropathic pain is due to Complex Regional Pain Syndrome (CRPS, Type I or Type II)
* NeP not due to trauma, and not peripheral pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Genk
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Pellenberg
  - Pfizer Investigational Site, Wilrijk
- Canada (4):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Denmark (2):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Hvidovre
- Finland (2):
  - Pfizer Investigational Site, HUS
  - Pfizer Investigational Site, Tampere
- Italy (3):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Montescano (PV)
  - Pfizer Investigational Site, Roma
- Netherlands (6):
  - Pfizer Investigational Site, Tilburg, North Brabant
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Kampen
  - Pfizer Investigational Site, Roosendaal
- Portugal (7):
  - Pfizer Investigational Site, Almada
  - Pfizer Investigational Site, Amadora
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Funchal
  - Pfizer Investigational Site, Guimarães
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Romania (2):
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Iași
- Sweden (3):
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Stockholm
- Switzerland (2):
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
- United Kingdom (4):
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Plymouth

REFERENCES:
- [Derived] van Seventer R, Serpell M, Bach FW, Morlion B, Zlateva G, Bushmakin AG, Cappelleri JC, Nimour M. Relationships between changes in pain severity and other patient-reported outcomes: an analysis in patients with posttraumatic peripheral neuropathic pain. Health Qual Life Outcomes. 2011 Mar 25;9:17. doi: 10.1186/1477-7525-9-17. PMID 21439051
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081064&StudyName=P4%20%28Pregabalin%20for%20Peripheral%20Posttraumatic%20Pain%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2-week screening period and single-blind washout and placebo run-in phase followed by a 4-week randomized, dose adjustment, double-blind treatment phase
Groups:
- Single-Blind Placebo: All subjects received placebo capsules for the 2-week screening period, subjects were then randomized to placebo or pregabalin treatment.
- Double-Blind Pregabalin: Dose adjustment of 150 to 600 mg/day based on tolerability through Visit 5. During the 4-week randomized maintenance phase, subjects maintained the same dosing regimen achieved at the end of the dose adjustment phase until the end of Week 8 (Visit 7).
  At the completion of the dose maintenance phase, subjects tapered off study medication during a 1-week double-blind taper phase (pregabalin 150 to 300 mg/day).
- Double-Blind Placebo: Matching placebo through Visit 5. During the 4-week randomized maintenance phase, subjects continued matching placebo until the end of Week 8 (Visit 7) and the 1 week taper phase.
Period: Single-Blind
Arm/Group | Single-Blind Placebo | Double-Blind Pregabalin | Double-Blind Placebo
Started | 368 | 0 | 0
Received Treatment | 367 | 0 | 0
Completed | 254 | 0 | 0
Not Completed | 114 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Laboratory Abnormality | 5 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Other | 77 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0
Not completed — Did not receive treatment | 1 | 0 | 0
Period: Double-Blind
Arm/Group | Single-Blind Placebo | Double-Blind Pregabalin | Double-Blind Placebo
Started | 0 | 127 | 127
Completed | 0 | 96 | 98
Not Completed | 0 | 31 | 29
Not completed — Adverse Event | 0 | 25 | 9
Not completed — Lack of Efficacy | 0 | 2 | 12
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Laboratory Abnormality | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Dose adjustment of 150 to 600 mg/day based on tolerability through Visit 5. During the 4-week randomized maintenance phase, subjects maintained the same dosing regimen achieved at the end of the dose adjustment phase until the end of Week 8 (Visit 7).
  At the completion of the dose maintenance phase, subjects tapered off study medication during a 1-week double-blind taper phase (pregabalin 150 to 300 mg/day).
- Placebo: Matching placebo through Visit 5. During the 4-week randomized maintenance phase, subjects continued matching placebo until the end of Week 8 (Visit 7) and the 1 week taper phase.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 127 | 127 | 254
Age, Customized [Number; unit: participants]
  18-44 years | 38 | 42 | 80
  45-64 years | 60 | 60 | 120
  ≥65 years | 29 | 25 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 52 | 129
  Male | 50 | 75 | 125

OUTCOME MEASURES:

1. Primary Outcome: Weekly Mean Pain Score at End of Treatment (Week 8) From Daily Pain Diary
Description: Daily Pain Diary scale : mean score from 11-point numerical scale of pain; range: 0 (no pain) to 10 (worst possible pain). Endpoint weekly mean pain score: mean of the last 7 available pain scores from a daily pain diary during double blind treatment.
Time Frame: each day of Week 8
Population: Full Analysis Set (FAS): all randomized subjects who received >= 1 dose study drug & have post-randomization efficacy data. Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 125
score on a scale | 4.61 (0.18) | 5.23 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; The study is powered to detect a clinically significant difference of 1 between treatment groups in the weekly mean pain score. Null hypothesis was that there was no difference in weekly mean pain scores between pregabalin and placebo; Test type: Superiority or Other; p = 0.010, ANCOVA; ANCOVA adjusted for treatment group, baseline mean pain score and pooled country; Mean Difference (Final Values) = -0.62, 95% CI [-1.09 to -0.15], Standard Error of Mean 0.24

2. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Anxiety Score
Description: Hospital Anxiety and Depression Scale Anxiety Score (HADS-A) consists of 7 items that are assessed by a score of 0 = no anxiety to 3 = severe feeling of anxiety. The anxiety subscale determines a state of generalized anxiety (including anxious mood, restlessness, anxious thoughts, panic attacks). Score range = 0 to 21; higher scores indicate a greater intensity of anxiety
Time Frame: Week 8
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 124 | 124
score on scale | 6.52 (0.29) | 7.36 (0.29)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.031, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -0.84, 95% CI [-1.60 to -0.08], Standard Error of Mean 0.39

3. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Depression Score
Description: Hospital Anxiety and Depression Scale Depression Score (HADS-D) consists of 7 items that are assessed by a score of 0 = no depression to 3 = severe feeling of depression. The depression subscale focuses on the state of lost interest and diminished pleasure response ("lowering of hedonic tone"). Score range = 0 to 21; higher scores indicate a greater intensity of depression
Time Frame: Week 8
Population: FAS LOCF
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 124 | 124
score on scale | 5.23 (0.24) | 6.20 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -0.97, 95% CI [-1.61 to -0.33], Standard Error of Mean 0.32

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Anxiety Score - FAS Subset With Moderate/Severe Baseline Scores
Description: as for outcome 2
Time Frame: Week 8
Population: Subset of subjects from the FAS who had moderate/severe baseline anxiety scores. LOCF.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 32 | 41
score on scale | 9.94 (0.77) | 11.63 (0.72)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.099, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -1.68, 95% CI [-3.69 to 0.32], Standard Error of Mean 1.00

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Depression Score - FAS Subset With Moderate/Severe Baseline Scores
Description: Hospital Anxiety and Depression Scale (HADS-D) consists of 7 items that are assessed by a score of 0 = no depression to 3 = severe feeling of depression. The depression subscale focuses on the state of lost interest and diminished pleasure response (lowering of hedonic tone). Score range = 0 to 21; higher scores indicate a greater intensity of depression
Time Frame: Week 8
Population: Subset of subjects from the FAS who had moderate/severe baseline depression scores. LOCF.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 17 | 23
score on scale | 12.04 (0.79) | 11.80 (0.79)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.819, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = 0.24, 95% CI [-1.87 to 2.34], Standard Error of Mean 1.03

6. Secondary Outcome: Weekly Mean Pain Score From Daily Pain Diary
Description: Daily Pain Diary scale : mean score from 11-point numerical scale of pain; range:0 (no pain) to 10 (worst possible pain). Mean of scores available for each week.
Time Frame: Baseline through Week 8
Population: FAS. Number of subjects with evaluable data: (n = pregabalin, placebo), respectively
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on scale
  Week 1 (n=125, 125) | 5.54 (0.11) | 5.79 (0.11)
  Week 2 (n=121, 119) | 5.37 (0.13) | 5.64 (0.13)
  Week 3 (n=113, 116) | 4.91 (0.15) | 5.44 (0.15)
  Week 4 (n=108, 108) | 4.95 (0.15) | 5.27 (0.15)
  Week 5 (n=106, 104) | 4.80 (0.16) | 5.26 (0.16)
  Week 6 (n=104, 101) | 4.76 (0.16) | 5.34 (0.16)
  Week 7 (n=99, 99) | 4.74 (0.18) | 5.26 (0.18)
  Week 8 (n=97, 97) | 4.64 (0.18) | 5.24 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.26, 95% CI [-0.56 to 0.05], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2: FAS; Test type: Superiority or Other; p = 0.150, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.26, 95% CI [-0.62 to 0.10], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3: FAS; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.53, 95% CI [-0.93 to -0.13], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4: FAS; Test type: Superiority or Other; p = 0.137, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.32, 95% CI [-0.74 to 0.10], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5: FAS; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.46, 95% CI [-0.90 to -0.02], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6: FAS; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.59, 95% CI [-1.03 to -0.15], Standard Error of Mean 0.22
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7: FAS; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.53, 95% CI [-1.01 to -0.04], Standard Error of Mean 0.25
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8: FAS; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; Repeated Measures Mixed Models. Adjusted for treatment, week, baseline pain score, pooled country and treatment-week; Mean Difference (Final Values) = -0.60, 95% CI [-1.10 to -0.10], Standard Error of Mean 0.25

7. Secondary Outcome: Number of Subjects With 30% and 50% Response in Weekly Mean Daily Pain Rating Score (DPRS) From Baseline Until Endpoint (Week 8)
Description: Based on weekly mean daily pain rating score (DPRS), responders were defined as subjects with a >= 30% and >=50% reduction in weekly mean scores from baseline until endpoint (Week 8). Endpoint was calculated as the mean of the last 7 available pain scores from the daily pain diary while in the double-blind treatment phase.
Time Frame: Baseline, Week 8
Population: FAS, LOCF.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 125
participants
  30% Responder | 50 | 32
  50% Responder | 30 | 18
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; 30% responder; Test type: Superiority or Other; p = 0.032, Regression, Logistic; logstic regression adjusted for treatment group, baseline pain score and pooled country; Odds Ratio (OR) = 1.84, 95% CI [1.05 to 3.21]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; 50% responder; Test type: Superiority or Other; p = 0.088, Regression, Logistic; logstic regression adjusted for treatment group, baseline pain score and pooled country; Odds Ratio (OR) = 1.78, 95% CI [0.92 to 3.46]

8. Secondary Outcome: Weekly Mean Sleep Interference Score
Description: 11-point numerical scale with which the patient describes pain interference with sleep over past 24 hours; range: 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep). Endpoint weekly mean score: mean of last 7 available scores from daily sleep interference diary during double-blind treatment.
Time Frame: Week 8
Population: FAS, LOCF
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 125
score on scale | 2.93 (0.17) | 3.73 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -0.79, 95% CI [-1.25 to -0.34], Standard Error of Mean 0.23

9. Secondary Outcome: Medical Outcome Study (MOS) Sleep Subscales
Description: Medical Outcome Study (MOS) is a patient-rated questionnaire consisting of 12 items that assess key constructs of sleep (7 subscales as well as a 9-item overall sleep problems index. MOS-Sleep Scale is scored from 0 to 100. A higher score indicates more disturbance.
Time Frame: Week 8
Population: FAS, LOCF. Number of subjects with evaluable data (n = pregabalin, placebo), respectively.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on a scale
  Sleep Disturbance (n=117, 118) | 35.73 (1.96) | 46.45 (1.94)
  Snoring (n=111, 118) | 38.92 (2.04) | 37.87 (1.97)
  Awaken Short of Breath/Headache (n= 118, 117) | 14.71 (2.14) | 20.66 (2.13)
  Sleep Quantity (n=117, 118) | 6.39 (0.32) | 6.48 (0.32)
  Sleep Adequacy (n=119, 119) | 55.25 (2.44) | 44.61 (2.43)
  Somnolence (n=116, 114) | 34.64 (1.75) | 32.33 (1.77)
  Sleep Problems Index-6 (n=112, 111) | 42.20 (1.96) | 51.72 (1.97)
  Sleep problems Index-9 (n=111, 107) | 35.43 (1.49) | 42.98 (1.52)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Sleep Disturbance; Test type: Superiority or Other; p = 0.000, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -10.72, 95% CI [-15.89 to -5.55], Standard Error of Mean 2.62
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Snoring; Test type: Superiority or Other; p = 0.700, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = 1.05, 95% CI [-4.30 to 6.40], Standard Error of Mean 2.71
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Awaken Short of Breath/Headache; Test type: Superiority or Other; p = 0.040, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -5.95, 95% CI [-11.62 to -0.28], Standard Error of Mean 2.88
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Sleep Quantity; Test type: Superiority or Other; p = 0.846, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -0.08, 95% CI [-0.92 to 0.76], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Sleep Adequacy; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = 10.63, 95% CI [4.19 to 17.07], Standard Error of Mean 3.27
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Somnolence; Test type: Superiority or Other; p = 0.324, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = 2.31, 95% CI [-2.30 to 6.92], Standard Error of Mean 2.34
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Sleep Problems Index-6; Test type: Superiority or Other; p = 0.000, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -9.52, 95% CI [-14.71 to -4.33], Standard Error of Mean 2.63
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Sleep Problems Index-9; Test type: Superiority or Other; p = 0.000, ANCOVA; ANCOVA adjusted for treatment group, baseline score and pooled country; Mean Difference (Final Values) = -7.54, 95% CI [-11.52 to -3.56], Standard Error of Mean 2.02

10. Secondary Outcome: Medical Outcome Study (MOS) Optimal Sleep
Description: Number of subjects responding to have had optimal sleep. Optimal sleep is 1 item in the Medical Outcome Study (MOS)sleep scale, a patient-reported measure consisting of twelve items that assess the key constructs of sleep. Subjects were asked to recall sleep-related activities over the past week.
Time Frame: Week 8
Population: FAS, LOCF.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 117 | 119
participants | 58 | 45
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.267, Regression, Logistic; Logistic regression adjusted for treatment group, baseline score and pooled country; Odds Ratio (OR) = 1.42, 95% CI [0.76 to 2.64]

11. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC): a patient-rated instrument that measures change in patient's overall status on a 7-point scale; range: 1 Very Much Improved to 7 Very Much Worse.
Time Frame: Week 8
Population: FAS, LOCF
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  very much improved | 13 | 6
  much improved | 27 | 22
  minimally improved | 41 | 26
  no change | 30 | 52
  minimally worse | 3 | 10
  much worse | 3 | 7
  very much worse | 3 | 2

12. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: Clinical Global Impression of Change (CGIC): clinician's judgment of overall change in the patient's condition over a defined period on a 7-point scale; range: 1 Very Much Improved to 7 Very Much Worse.
Time Frame: Week 8
Population: FAS, LOCF
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  very much improved | 11 | 6
  much improved | 33 | 18
  minimally improved | 36 | 26
  no change | 33 | 61
  minimally worse | 5 | 9
  much worse | 4 | 3
  very much worse | 1 | 1

13. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Impact of Current Pain Medication
Description: Pain Treatment Satisfaction Scale (PTSS); Impact of Current Pain Medication: measure of patient satisfaction with treatment for acute or chronic pain. Response range: 1 (strongly agree) to 5 (strongly disagree). Mean scores were calculated and transformed onto a scale of 0-100, range: 0 = worst possible satisfaction to 100 = best possible satisfaction with pain treatment.
Time Frame: Screening, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 127
score on a scale
  Screening (n=113, 113) | 54.53 (27.60) | 53.60 (26.07)
  End of Treatment (Week 8) (n=122, 121) | 52.64 (31.87) | 42.56 (32.52)

14. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Satisfaction With Current Pain Medication
Description: Pain Treatment Satisfaction Scale (PTSS); Satisfaction with Current Pain Medication: measure of patient satisfaction with treatment for acute or chronic pain. Response range:1 (strongly agree) to 5 (strongly disagree). Mean scores were calculated and transformed onto a scale of 0-100, range: 0 = worst possible satisfaction to 100 = best possible satisfaction with pain treatment.
Time Frame: Screening, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 122 | 121
score on scale
  Screening (n=112, 110) | 50.33 (20.85) | 51.05 (20.52)
  Week 8 (n=122, 121) | 62.36 (22.22) | 54.15 (22.78)

15. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Medication Characteristics
Description: Pain Treatment Satisfaction Scale (PTSS); Medication Characteristics: measure of patient satisfaction with treatment for acute or chronic pain. Response range: 1 (strongly agree) to 5 (strongly disagree). Mean scores were calculated and transformed onto a scale of 0-100, range: 0 = worst possible satisfaction to 100 = best possible satisfaction with pain treatment.
Time Frame: Screening, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 127
score on scale
  Screening (n=112, 110) | 57.44 (21.84) | 59.39 (22.21)
  End of Treatment (Week 8) (n=122, 121) | 71.52 (19.58) | 70.39 (21.00)

16. Secondary Outcome: Pain Treatment Satisfaction Scale (PTSS): Efficacy
Description: Pain Treatment Satisfaction Scale (PTSS); Efficacy: measure of patient satisfaction with treatment for acute or chronic pain. Response range: 1 (strongly agree) to 5 (strongly disagree). Mean scores were calculated and transformed onto a scale of 0-100, range: 0 = worst possible satisfaction to 100 = best possible satisfaction with pain treatment.
Time Frame: Screening, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 127
score on scale
  Screening (n=112, 110) | 43.23 (24.06) | 42.73 (23.98)
  End of Treatment (Week 8) (n=122, 121) | 53.21 (30.63) | 37.88 (32.61)

17. Secondary Outcome: Modified Brief Pain Inventory Short Form (m-BPI-sf)
Description: Modified Brief Pain Inventory Short Form (m-BPI-sf): self-administered questionnaire to assess severity of pain (measured by 4 items)and impact of pain on daily functions (measured by 7 items)in past 24 hours. Items are rated on an 11-point scale ranging from 0 to 10, with higher scores indicating greater pain and/or interference due to pain.
Time Frame: Baseline, Week 8
Population: Baseline; FAS, LOCF. Number of subjects with evaluable data: (n = pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on a scale
  pain interference index Baseline (n=125, 126) | 4.57 (2.11) | 4.69 (2.36)
  pain interference index Week 8 (n=120, 121) | 3.31 (2.41) | 4.17 (2.49)
  pain severity index Baseline (n= 122, 125) | 5.36 (1.71) | 5.72 (2.04)
  pain severity index Week 8 (n=120, 120) | 4.20 (2.35) | 5.21 (2.42)

18. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI) Total Intensity Score
Description: Neuropathic Pain Symptom Inventory (NPSI) includes 10 descriptors (scale 0-10) of different pain symptoms & 2 temporal items assessing the duration of spontaneous ongoing and paroxysmal pain. A total intensity score is calculated by sub grouping the questions into five pain dimensions, summing the five sub groups, and converting into a percentage.
Time Frame: Week 8
Population: FAS. Number of subjects with a non-missing NPSI Total Intensity Score at Baseline and Week 8 (using LOCF) is 100, 106 for pregabalin, placebo respectively.
Measure: Least Squares Mean (Standard Error); unit: percentage score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
percentage score on scale | 33.29 (1.68) | 37.12 (1.66)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.090, ANCOVA; Mean Difference (Final Values) = -3.84, 95% CI [-8.28 to 0.61], Standard Error of Mean 2.25

19. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Reasoning
Description: The number of subjects' responses to each of the 6 questions on the Medical Outcome Study Cognitive (MOS-Cog) subscale were summarized at baseline and Week 8. Category range: all of the time to none of the time. No formal statistical modeling was used.
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 120, 121 for pregabalin, placebo respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  Baseline: All of the Time | 5 | 1
  Baseline: Most of the Time | 6 | 15
  Baseline: A Good Bit of the Time | 5 | 15
  Baseline: Some of the Time | 20 | 25
  Baseline: A Little of the Time | 42 | 27
  Baseline: None of the Time | 48 | 43
  Week 8: All of the Time | 3 | 4
  Week 8: Most of the Time | 10 | 5
  Week 8: A Good Bit of the Time | 11 | 13
  Week 8: Some of the Time | 23 | 27
  Week 8: A Little of the Time | 32 | 30
  Week 8: None of the Time | 41 | 42

20. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Concentration
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 120, 121 for pregabalin, placebo respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  Baseline: All of the Time | 4 | 4
  Baseline: Most of the Time | 8 | 14
  Baseline: A Good Bit of the Time | 13 | 14
  Baseline: Some of the Time | 27 | 29
  Baseline: A Little of the Time | 33 | 26
  Baseline: None of the Time | 41 | 39
  Week 8: All of the Time | 3 | 7
  Week 8: Most of the Time | 12 | 5
  Week 8: A Good Bit of the Time | 14 | 16
  Week 8: Some of the Time | 26 | 27
  Week 8: A Little of the Time | 27 | 33
  Week 8: None of the Time | 38 | 33

21. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Confusion
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 119, 121 for pregabalin, placebo respectively.
Measure: Number; unit: particpants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
particpants
  Baseline: All of the Time | 2 | 6
  Baseline: Most of the Time | 8 | 12
  Baseline: A Good Bit of the Time | 6 | 7
  Baseline: Some of the Time | 22 | 15
  Baseline: A Little of the Time | 23 | 35
  Baseline: None of the Time | 64 | 51
  Week 8: All of the Time | 1 | 3
  Week 8: Most of the Time | 9 | 11
  Week 8: A Good Bit of the Time | 9 | 6
  Week 8: Some of the Time | 26 | 23
  Week 8: A Little of the Time | 22 | 27
  Week 8: None of the Time | 52 | 51

22. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Memory
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 120, 121 for pregabalin, placebo respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  Baseline: All of the Time | 7 | 10
  Baseline: Most of the Time | 7 | 14
  Baseline: A Good Bit of the Time | 6 | 8
  Baseline: Some of the Time | 40 | 23
  Baseline: A Little of the Time | 30 | 33
  Baseline: None of the Time | 36 | 38
  Week 8: All of the Time | 3 | 9
  Week 8: Most of the Time | 11 | 7
  Week 8: A Good Bit of Time | 13 | 11
  Week 8: Some of the Time | 28 | 31
  Week 8: A Little of the Time | 36 | 35
  Week 8: None of the Time | 29 | 28

23. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Attention
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 120, 121 for pregabalin, placebo respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  Baseline: All of the Time | 5 | 3
  Baseline: Most of the Time | 3 | 16
  Baseline: A Good Bit of Time | 13 | 14
  Baseline: Some of the Time | 24 | 23
  Baseline: A Little of the Time | 39 | 23
  Baseline: None of the Time | 42 | 47
  Week 8: All of the Time | 4 | 5
  Week 8: Most of the Time | 10 | 7
  Week 8: A Good Bit of Time | 8 | 13
  Week 8: Some of the Time | 22 | 26
  Week 8: A Little of the Time | 34 | 34
  Week 8: None of the Time | 42 | 36

24. Secondary Outcome: Medical Outcome Study Cognitive Subscale (MOS-Cog); Thinking
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: FAS, LOCF. The number of subjects that answered the question at Week 8 is 120, 121 for pregabalin, placebo respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
participants
  Baseline: All of the Time | 2 | 1
  Baseline: Most of the Time | 6 | 9
  Baseline: A Good Bit of Time | 3 | 6
  Baseline: Some of the Time | 31 | 27
  Baseline: A Little of the Time | 33 | 36
  Baseline: None of the Time | 51 | 45
  Week 8: All of the Time | 4 | 6
  Week 8: Most of the Time | 6 | 9
  Week 8: A Good Bit of Time | 12 | 6
  Week 8: Some of the Time | 28 | 22
  Week 8: A Little of the Time | 31 | 31
  Week 8: None of the Time | 39 | 47

25. Secondary Outcome: Davidson Trauma Scale (DTS): Severity
Description: Self-rated instrument to measure symptom severity and treatment outcome in post traumatic stress disorder (PTSD). Scale of 17 PTSD symptoms over previous week; frequency scale: 0 (not at all) to 4 (every day), and severity 0 (not at all distressing) to 4(extremely distressing). The total Davidson Trauma Scale score ranges from 0 to 136.
Time Frame: Baseline, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data: (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on a scale
  Baseline (n=116, 118) | 15.55 (14.16) | 17.83 (16.94)
  Week 8 (n=112, 113) | 11.71 (13.77) | 15.43 (16.91)

26. Secondary Outcome: Davidson Trauma Scale (DTS): Frequency
Description: as for outcome 25
Time Frame: Baseline, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data: (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on scale
  Baseline (n=124, 124) | 18.27 (13.98) | 20.90 (15.11)
  Week 8 (n=118, 120) | 14.16 (12.67) | 18.47 (15.51)

27. Secondary Outcome: Davidson Trauma Scale (DTS): Total Score
Description: as for outcome 25
Time Frame: Baseline, Week 8
Population: FAS, LOCF. Number of subjects with evaluable data: (n=pregabalin, placebo), respectively.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 126 | 126
score on scale
  Baseline (n=116, 118) | 34.57 (27.56) | 38.76 (31.55)
  Week 8 (n=112, 113) | 26.18 (26.09) | 33.62 (31.65)

ADVERSE EVENTS:
Arm/Group | Single-Blind Placebo | Double-Blind Pregabalin | Double-Blind Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 4 | 2
Other Adverse Events (participants affected / at risk) | 77 | 109 | 73
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Single-Blind Placebo | Double-Blind Pregabalin | Double-Blind Placebo
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/367 | 1/127 | 0/127
Back pain (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Viral infection (Infections and infestations) | 1/367 | 1/127 | 0/127
Fall (Injury, poisoning and procedural complications) | 0/367 | 0/127 | 1/127
Skin laceration (Injury, poisoning and procedural complications) | 0/367 | 0/127 | 1/127
Foot fracture (Injury, poisoning and procedural complications) | 0/367 | 0/127 | 1/127
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0/367 | 1/127 | 0/127
Tremor (Nervous system disorders) | 0/367 | 1/127 | 0/127
Confusional state (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Accidental Over Dose (Injury, poisoning and procedural complications) | 1/367 | 0/127 | 1/127
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Single-Blind Placebo | Double-Blind Pregabalin | Double-Blind Placebo
Leukopenia (Blood and lymphatic system disorders) | 0/367 | 1/127 | 0/127
Blood calcium increased (Investigations) | 0/367 | 1/127 | 0/127
Thrombocytopenia (Blood and lymphatic system disorders) | 0/367 | 1/127 | 0/127
Blood cholesterol increased (Investigations) | 0/367 | 1/127 | 0/127
Palpitations (Cardiac disorders) | 1/367 | 0/127 | 0/127
Hypoacusis (Ear and labyrinth disorders) | 0/367 | 0/127 | 1/127
Vertigo (Ear and labyrinth disorders) | 0/367 | 4/127 | 1/127
Goitre (Endocrine disorders) | 0/367 | 1/127 | 0/127
Hyperthyroidism (Endocrine disorders) | 0/367 | 0/127 | 1/127
Hypothyroidism (Endocrine disorders) | 0/367 | 0/127 | 1/127
Thyroid disorder (Endocrine disorders) | 0/367 | 0/127 | 1/127
Abnormal sensation in eye (Eye disorders) | 0/367 | 1/127 | 0/127
Altered visual depth perception (Eye disorders) | 0/367 | 1/127 | 0/127
Blepharospasm (Eye disorders) | 0/367 | 0/127 | 1/127
Diplopia (Eye disorders) | 1/367 | 0/127 | 0/127
Vision blurred (Eye disorders) | 3/367 | 8/127 | 3/127
Visual acuity reduced (Eye disorders) | 0/367 | 0/127 | 1/127
Abdominal discomfort (Gastrointestinal disorders) | 1/367 | 1/127 | 1/127
Abdominal pain upper (Gastrointestinal disorders) | 1/367 | 2/127 | 2/127
Constipation (Gastrointestinal disorders) | 1/367 | 9/127 | 4/127
Diarrhoea (Gastrointestinal disorders) | 5/367 | 5/127 | 5/127
Dry mouth (Gastrointestinal disorders) | 5/367 | 14/127 | 6/127
Dyspepsia (Gastrointestinal disorders) | 2/367 | 2/127 | 0/127
Flatulence (Gastrointestinal disorders) | 1/367 | 2/127 | 0/127
Frequent bowel movements (Gastrointestinal disorders) | 1/367 | 1/127 | 0/127
Gastric disorder (Gastrointestinal disorders) | 0/367 | 0/127 | 1/127
Gastritis (Gastrointestinal disorders) | 0/367 | 0/127 | 1/127
Haemorrhoids (Gastrointestinal disorders) | 0/367 | 1/127 | 0/127
Hyperchlorhydria (Gastrointestinal disorders) | 0/367 | 0/127 | 1/127
Hypoaesthesia oral (Gastrointestinal disorders) | 0/367 | 0/127 | 2/127
Irritable bowel syndrome (Gastrointestinal disorders) | 0/367 | 1/127 | 0/127
Nausea (Gastrointestinal disorders) | 8/367 | 12/127 | 8/127
Toothache (Gastrointestinal disorders) | 0/367 | 1/127 | 0/127
Vomiting (Gastrointestinal disorders) | 1/367 | 4/127 | 2/127
Asthenia (General disorders) | 0/367 | 2/127 | 0/127
Chest discomfort (General disorders) | 0/367 | 1/127 | 0/127
Chest pain (General disorders) | 3/367 | 0/127 | 0/127
Fatigue (General disorders) | 4/367 | 15/127 | 10/127
Feeling abnormal (General disorders) | 0/367 | 1/127 | 0/127
Feeling drunk (General disorders) | 0/367 | 5/127 | 0/127
Feeling hot (General disorders) | 0/367 | 0/127 | 1/127
Feeling jittery (General disorders) | 0/367 | 1/127 | 0/127
Gait disturbance (General disorders) | 0/367 | 1/127 | 0/127
Hunger (General disorders) | 1/367 | 0/127 | 0/127
Influenza like illness (General disorders) | 1/367 | 0/127 | 0/127
Irritatibility (General disorders) | 0/367 | 0/127 | 2/127
Localised oedema (General disorders) | 0/367 | 1/127 | 0/127
Malaise (General disorders) | 0/367 | 0/127 | 1/127
Mucosal dryness (General disorders) | 1/367 | 1/127 | 0/127
Oedema peripheral (General disorders) | 1/367 | 9/127 | 3/127
Pain (General disorders) | 3/367 | 5/127 | 0/127
Thirst (General disorders) | 0/367 | 2/127 | 2/127
Hypersensitivity (Immune system disorders) | 0/367 | 1/127 | 0/127
Bronchitis (Infections and infestations) | 0/367 | 2/127 | 0/127
Cystitis (Infections and infestations) | 0/367 | 0/127 | 1/127
Gastroenteritis (Infections and infestations) | 1/367 | 1/127 | 0/127
Herpes simplex (Infections and infestations) | 1/367 | 1/127 | 0/127
Herpes zoster (Infections and infestations) | 0/367 | 1/127 | 0/127
Infulenza (Infections and infestations) | 2/367 | 3/127 | 2/127
Lower respiratory tract infection (Infections and infestations) | 0/367 | 2/127 | 0/127
Lung infection (Infections and infestations) | 1/367 | 0/127 | 0/127
Nasopharyngitis (Infections and infestations) | 2/367 | 1/127 | 3/127
Pharyngitis (Infections and infestations) | 1/367 | 2/127 | 0/127
Pneumonia (Infections and infestations) | 0/367 | 0/127 | 1/127
Respiratory tract infection (Infections and infestations) | 0/367 | 1/127 | 0/127
Schistomosomiasis cutaneous (Infections and infestations) | 0/367 | 1/127 | 0/127
Sinusitis (Infections and infestations) | 0/367 | 0/127 | 1/127
Skin infection (Infections and infestations) | 1/367 | 0/127 | 1/127
Tooth infection (Infections and infestations) | 0/367 | 0/127 | 1/127
Upper respiratory tract infection (Infections and infestations) | 0/367 | 3/127 | 0/127
Urinary tract infection (Infections and infestations) | 0/367 | 1/127 | 0/127
Viral infection (Infections and infestations) | 1/367 | 0/127 | 1/127
Viral upper respiratory tract infection (Infections and infestations) | 0/367 | 1/127 | 1/127
Accidental overdose (Injury, poisoning and procedural complications) | 0/367 | 1/127 | 0/127
Arthropod bite (Injury, poisoning and procedural complications) | 0/367 | 0/127 | 1/127
Fall (Injury, poisoning and procedural complications) | 1/367 | 2/127 | 3/127
Joint sprain (Injury, poisoning and procedural complications) | 0/367 | 1/127 | 0/127
Muscle strain (Injury, poisoning and procedural complications) | 0/367 | 1/127 | 0/127
Skeletal injury (Injury, poisoning and procedural complications) | 0/367 | 0/127 | 1/127
Skin laceration (Injury, poisoning and procedural complications) | 0/367 | 2/127 | 0/127
Blood glucose increased (Investigations) | 0/367 | 0/127 | 1/127
Blood pressure systolic increased (Investigations) | 0/367 | 0/127 | 1/127
Blood thyroid stimulating hormone increased (Investigations) | 0/367 | 1/127 | 1/127
Blood triglycerides decreased (Investigations) | 0/367 | 0/127 | 1/127
Blood triglycerides increased (Investigations) | 0/367 | 0/127 | 2/127
Creatinine renal clearance decreased (Investigations) | 2/367 | 0/127 | 0/127
Drug screen positive (Investigations) | 1/367 | 0/127 | 0/127
Haemoglobin increased (Investigations) | 0/367 | 0/127 | 1/127
Neutrophil count increased (Investigations) | 0/367 | 0/127 | 1/127
Wieght increased (Investigations) | 1/367 | 5/127 | 2/127
Fluid retention (Metabolism and nutrition disorders) | 0/367 | 1/127 | 0/127
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/367 | 1/127 | 1/127
Increased appetite (Metabolism and nutrition disorders) | 2/367 | 2/127 | 3/127
Polydipsia (Metabolism and nutrition disorders) | 1/367 | 0/127 | 0/127
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/367 | 3/127 | 2/127
Arthritis (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Arthropathy (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Back pain (Musculoskeletal and connective tissue disorders) | 2/367 | 1/127 | 2/127
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1/367 | 1/127 | 0/127
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/367 | 1/127 | 0/127
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/367 | 1/127 | 1/127
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/367 | 1/127 | 0/127
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/367 | 1/127 | 0/127
Myalgia (Musculoskeletal and connective tissue disorders) | 1/367 | 0/127 | 1/127
Neck pain (Musculoskeletal and connective tissue disorders) | 0/367 | 0/127 | 1/127
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/367 | 1/127 | 2/127
Ataxia (Nervous system disorders) | 0/367 | 1/127 | 0/127
Balance disorder (Nervous system disorders) | 0/367 | 4/127 | 0/127
Coordination abnormal (Nervous system disorders) | 0/367 | 1/127 | 0/127
Crying (Nervous system disorders) | 1/367 | 0/127 | 0/127
Disturbance in attention (Nervous system disorders) | 1/367 | 9/127 | 4/127
Dizziness (Nervous system disorders) | 10/367 | 55/127 | 12/127
Dysaesthesia (Nervous system disorders) | 0/367 | 1/127 | 0/127
Dysarthria (Nervous system disorders) | 0/367 | 2/127 | 0/127
Dyskinesia (Nervous system disorders) | 0/367 | 1/127 | 0/127
Formication (Nervous system disorders) | 1/367 | 1/127 | 1/127
Head discomfort (Nervous system disorders) | 1/367 | 1/127 | 0/127
Headache (Nervous system disorders) | 14/367 | 15/127 | 14/127
Hypoaesthesia (Nervous system disorders) | 0/367 | 1/127 | 0/127
Memory impairment (Nervous system disorders) | 0/367 | 4/127 | 3/127
Mental impairment (Nervous system disorders) | 0/367 | 2/127 | 0/127
Migraine (Nervous system disorders) | 0/367 | 1/127 | 0/127
Neuralgia (Nervous system disorders) | 1/367 | 5/127 | 2/127
Paraesthesia (Nervous system disorders) | 2/367 | 3/127 | 0/127
Sciatica (Nervous system disorders) | 1/367 | 2/127 | 0/127
Somnolence (Nervous system disorders) | 3/367 | 20/127 | 8/127
Speech disorder (Nervous system disorders) | 0/367 | 1/127 | 0/127
Syncope (Nervous system disorders) | 0/367 | 1/127 | 0/127
Tension headache (Nervous system disorders) | 0/367 | 0/127 | 1/127
Tremor (Nervous system disorders) | 0/367 | 1/127 | 1/127
Abnormal dreams (Psychiatric disorders) | 0/367 | 2/127 | 0/127
Agitation (Psychiatric disorders) | 1/367 | 1/127 | 0/127
Anxiety (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Daydreaming (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Deja vu (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Depression (Psychiatric disorders) | 2/367 | 1/127 | 0/127
Disinhibition (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Disorientation (Psychiatric disorders) | 0/367 | 2/127 | 0/127
Dissociation (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Dyssomnia (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Emotional disorder (Psychiatric disorders) | 0/367 | 0/127 | 1/127
Encopresis (Psychiatric disorders) | 1/367 | 1/127 | 0/127
Euphoric (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Insomnia (Psychiatric disorders) | 1/367 | 1/127 | 6/127
Libido decreased (Psychiatric disorders) | 0/367 | 0/127 | 1/127
Mood altered (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Morose (Psychiatric disorders) | 0/367 | 0/127 | 1/127
Nervousness (Psychiatric disorders) | 0/367 | 0/127 | 1/127
Nightmare (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Alopecia (Skin and subcutaneous tissue disorders) | 1/367 | 1/127 | 0/127
Restlessness (Psychiatric disorders) | 0/367 | 1/127 | 1/127
Sleep disorder (Psychiatric disorders) | 0/367 | 0/127 | 2/127
Tic (Psychiatric disorders) | 0/367 | 1/127 | 0/127
Haematuria (Renal and urinary disorders) | 0/367 | 1/127 | 0/127
Polyuria (Renal and urinary disorders) | 2/367 | 1/127 | 0/127
Urinary retention (Renal and urinary disorders) | 0/367 | 0/127 | 1/127
Dysmenorrhoea (Reproductive system and breast disorders) | 0/367 | 1/127 | 0/127
Sexual dysfunction (Reproductive system and breast disorders) | 0/367 | 0/127 | 1/127
Cough (Respiratory, thoracic and mediastinal disorders) | 0/367 | 0/127 | 1/127
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/367 | 1/127 | 0/127
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0/367 | 1/127 | 2/127
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0/367 | 0/127 | 1/127
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 0/367 | 1/127 | 1/127
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/367 | 1/127 | 0/127
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/367 | 0/127 | 1/127
Acne (Skin and subcutaneous tissue disorders) | 0/367 | 0/127 | 1/127
Dermatitis (Skin and subcutaneous tissue disorders) | 0/367 | 1/127 | 0/127
Dry skin (Skin and subcutaneous tissue disorders) | 0/367 | 3/127 | 1/127
Erythema (Skin and subcutaneous tissue disorders) | 0/367 | 2/127 | 0/127
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/367 | 4/127 | 1/127
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0/367 | 1/127 | 0/127
Night sweats (Skin and subcutaneous tissue disorders) | 1/367 | 0/127 | 2/127
Rash (Skin and subcutaneous tissue disorders) | 0/367 | 1/127 | 2/127
Rash pruritic (Skin and subcutaneous tissue disorders) | 0/367 | 0/127 | 2/127
Skin discolouration (Skin and subcutaneous tissue disorders) | 0/367 | 1/127 | 0/127
Breast prothesis implantation (Surgical and medical procedures) | 0/367 | 0/127 | 1/127
Hot flush (Vascular disorders) | 1/367 | 0/127 | 0/127
Hypertension (Vascular disorders) | 1/367 | 5/127 | 2/127
Hypotension (Vascular disorders) | 1/367 | 1/127 | 2/127
Thrombophlebitis superficial (Vascular disorders) | 0/367 | 1/127 | 0/127
Blood calcium decreased (Investigations) | 0/367 | 1/127 | 0/127
Adominal pain (Gastrointestinal disorders) | 1/367 | 1/127 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.